CLINICAL TRIAL: NCT00453037
Title: Effects of a Structured Education Program on Blood Pressure in Essential Hypertensive Patients and Effects of a Reminder Program for Physicians to Guide Optimal Therapy
Brief Title: Effects of a Structured Education Program on Blood Pressure in Essential Hypertensive Patients
Acronym: herzleben
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Medical University of Graz, Dept of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17019ex05-06
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Hypertension
Keywords: hypertension; self measurement of blood pressure; education program; life style
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group I (early intervention) (Active Comparator): We refer to the results of the DAFNE-study. This study showed the merits of an educational program in diabetics. In accordance to the protocol of DAFNE, we developed a design as follows: For each participating center patients are randomly assigned to two groups. Group I receives an early educational intervention at time of randomization, which should lead to better control of blood pressure after 6 months compared to the control group. The protocol design was chosen for proving an independent effect of the educational program despite optimal management by the GP. Group II is designated to receive the educational intervention 6 months after enrollment into the study.
  for further details please see brief description section
  Interventions: Behavioral: structured educational program
- delayed education (Other): delayed educational intervention
  for further details please see brief description section
  Interventions: Behavioral: participation in the educational program after 6 months

INTERVENTIONS:
Behavioral: structured educational program — structured education and evaluation of hypertensive patients in a design similar to the DAFNE study design. Behavioural intervention follows the Dusseldorf-educational program
  Other Names: educational program at time of inclusion; delayed educational program six moth later
  Arms: group I (early intervention)
Behavioral: participation in the educational program after 6 months — Control group consisting of patients randomly assigned to participate in the educational program 6 months later than the active group
  Arms: delayed education

SUMMARY:
The purpose of this study is to evaluate the effects of a structured educational program for hypertensive patients. The program was developed at the University of Dusseldorf, Germany. The contents of the program are as follows: teaching of the background of hypertension, techniques of self estimation of blood pressure, life style and dietary habits, some information concerning the different pharmacological properties to treat hypertension

DETAILED DESCRIPTION:
see brief description section

ELIGIBILITY:
Inclusion Criteria:

* Intellectual and physical ability to attend teaching program,
* Capability to do and document blood pressure self-measurement,
* Systolic blood pressure >160 and/or diastolic blood pressure >95 mmHg,
* At least 3 months of preexisting medicamentous anti-hypertensive treatment,
* 15% or higher risc in New Zealand Risc Scale

Exclusion Criteria:

* Failing inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure at 6 and 12 months of follow up following the educational process | 1 year

SECONDARY OUTCOMES:
morbidity on different cardiovascular and cerebrovascular diseases | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zweiker, MD AssocProf, Principal Investigator — Medical University Graz Dep of Internal Medicine; Div of Cardiology; Thomas R Pieber, MD AssocProf, Principal Investigator — Medical University Graz Dept of Internal Medicine Div of Diabetology
Locations (1):
- Medical University Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Perl S, Niederl E, Kos C, Mrak P, Ederer H, Rakovac I, Beck P, Kraler E, Stoff I, Klima G, Pieske BM, Pieber TR, Zweiker R. Randomized Evaluation of the Effectiveness of a Structured Educational Program for Patients With Essential Hypertension. Am J Hypertens. 2016 Jul;29(7):866-72. doi: 10.1093/ajh/hpv186. Epub 2015 Dec 7. PMID 26643687